CLINICAL TRIAL: NCT05845593
Title: An Open Label Multicenter Study to Assess the Relationship Between Data Obtained With the LuGENE® Multiparameter Transcriptomics Blood Test and Clinical and Standard Laboratory Features of Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Relationship Between Data Obtained With the LuGENE® Multiparameter Transcriptomics Blood Test and Clinical and Standard Laboratory Features of Patients With SLE (ReLATE)
Acronym: ReLATE
Status: Recruiting | Type: Observational
Sponsor: Ampel BioSolutions, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AMP-005
Record Dates: First submitted 2023-04-04; First posted 2023-05-06 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Future Research Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Adult male and female patients with a clinical diagnosis of SLE or incomplete lupus
  Interventions: Other: Decision Support Test

INTERVENTIONS:
Other: Decision Support Test — LuGENE®, a transcriptomic-based LDT, with standard evaluation of patients diagnosed with SLE

SUMMARY:
This is an open label study to determine the association of the data obtained with LuGENE®, a transcriptomic-based LDT, with standard evaluation of patients diagnosed with SLE, including clinical involvement, SLEDAI score, Physician Global Assessment (PGA) and standard laboratory measures, including ANA, anti-DNA, anti-RNP and complement components C3 and C4, as well as Patient Reported Outcomes capturing pain, fatigue and Health-Related Quality of Life. The test will be administered on one occasion to patients with a clinical diagnosis of lupus or incomplete lupus and clinical and laboratory features evaluated contemporaneously. This trial includes a pilot study of approximately 10 subjects from 2-3 sites to assess whether the delivery times of LuGENE® laboratory results do not exceed more than 7 business days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged at least 18 years old.
2. Capable of giving written consent on an IRB-approved Informed Consent Form prior to any study-specific evaluation
3. Have a clinical diagnosis of SLE determined by the examining physician or a diagnosis of incomplete lupus determined by the examining physician
4. On a stable SLE treatment regimen consisting of a stable dosage of medications for a period of at least 30 days prior to testing

Exclusion Criteria:

1. Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not related to SLE (i.e., diabetes, cardiovascular, pulmonary, hematologic, gastrointestinal, neurological, or infectious) which, in the opinion of the treating physician, could confound the results of the study or put the patient at undue risk
2. Have received intravenous glucocorticoids at a dosage of ≥ 500 mg daily within the past month
3. Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Baseline
4. Pregnant or lactating.
5. Recent participation in a clinical trial with an experimental agent in the past 6 weeks, or 5 half-lives of the study drug, whichever is longer
6. Any condition that in the opinion of the treating physician might interfere with the performance of the LuGENE® test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients with a clinical diagnosis of SLE or incomplete lupus
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-03-05 (Estimated)

PRIMARY OUTCOMES:
LuGENE clinical decision support relative to clinical disease activity | 16 months
  The primary endpoint is to determine the capacity of LuGENE® to support clinical decision making by Health Care Professionals (HCPs) providing care to lupus patients. This will be determined by comparing the data obtained with LuGENE®, a transcriptomic-based LDT, with standard evaluation of patients diagnosed with SLE, including clinical activity (SLEDAI score) Physician Global Assessment (PGA).
LuGENE clinical decision support relative to lab measures | 16 months
  The co-primary endpoint is to determine the capacity of LuGENE® to support clinical decision making by Health Care Professionals (HCPs) providing care to lupus patients. This will be determined by comparing the data obtained with LuGENE® with standard laboratory measures of lupus (ANA, anti-DNA, anti-RNP and complement components C3 and C4)
LuGENE clinical decision support relative to PROs | 16 months
  The co-primary endpoint is to determine the capacity of LuGENE® to support clinical decision making by Health Care Professionals (HCPs) providing care to lupus patients. This will be determined by comparing the data obtained with LuGENE with standard evaluation of patient reported outcomes using standard instruments capturing pain, fatigue and Health-Related Quality of Life.

SECONDARY OUTCOMES:
LuGENE score correlation to Immune Function with Biomarker endpoint: | 16 months
  The association of the LuGENE Score with Immune function in SLE patients using Biomarkers (Anti-DNA, anti-RNP, Complement C3/C4 levels).
LuGENE score correlation to Clinical Feature endpoint: | 16 months
  The association of the LuGENE Score with Clinical features of SLE using SLEDAI-2K with sub-domains, ACR/EULAR Lupus diagnostic criteria, Physician Global Assessment (PGA)
LuGENE score correlation to Quality of Life PROs endpoint: | 16 months
  The association of the LuGENE Score with Quality of Life measures using validated patient PROs (SF-36, fatigue by FACIT-F, Fatigue VAS, Pain VAS, Patient Global Assessment (PtGA))
LuGENE subset membership correlation to Immune Function with Biomarker endpoint: | 16 months
  The association of the LuGENE® determined subset membership with Immune function in SLE patients using Biomarkers (Anti-DNA, anti-RNP, Complement C3/C4 levels).
LuGENE subset membership correlation to Clinical Feature endpoint: | 16 months
  The association of the LuGENE® determined subset membership with Clinical features of SLE using SLEDAI-2K with sub-domains, ACR/EULAR Lupus diagnostic criteria, Physician Global Assessment (PGA)
LuGENE subset membership correlation to Quality of Life PROs endpoint: | 16 months
  The association of the LuGENE® determined subset membership with Quality of Life measures using validated patient PROs (SF-36, fatigue by FACIT-F, Fatigue VAS, Pain VAS, Patient Global Assessment (PtGA))
LuGENE profile correlation to Immune Function with Biomarker endpoint: | 16 months
  The association of the LuGENE® profile with Immune function in SLE patients using Biomarkers (Anti-DNA, anti-RNP, Complement C3/C4 levels).
LuGENE profile correlation to Clinical Feature endpoint: | 16 months
  The association of the LuGENE® profile with Clinical features of SLE using SLEDAI-2K with sub-domains, ACR/EULAR Lupus diagnostic criteria, Physician Global Assessment (PGA)
LuGENE profile correlation to Quality of Life PROs endpoint: | 16 months
  The association of the LuGENE® profile with Quality of Life measures using validated patient PROs (SF-36, fatigue by FACIT-F, Fatigue VAS, Pain VAS, Patient Global Assessment (PtGA))

OTHER OUTCOMES:
Physician use and satisfaction | 16 months
  Evaluate the patterns of physician use and opinion of value of LuGENE® using a focused questionnaire created for this trial

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Providence St. John's Health Center - Rheumatology, Santa Monica, California
  - Yale School of Medicine, New Haven, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Feinstein Institute for Medical Research, Manhasset, New York
  - The Hospital for Special Surgery, New York, New York
  - Arthritis and Osteoporosis Consultants of the Carolinas, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hubbard EL, Bachali P, Kingsmore KM, He Y, Catalina MD, Grammer AC, Lipsky PE. Analysis of transcriptomic features reveals molecular endotypes of SLE with clinical implications. Genome Med. 2023 Oct 16;15(1):84. doi: 10.1186/s13073-023-01237-9. PMID 37845772
- See also: Related Info — https://genomemedicine.biomedcentral.com/articles/10.1186/s13073-023-01237-9